CLINICAL TRIAL: NCT04024306
Title: Steroid-induced Diabetes Mellitus in Systemic Lupus Erythematosus (SLE) Patients
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: Assiut University (Other)
Responsible Party: Principal Investigator, Muhammad Abd-Erazek Ahmad, Assiut, Egypt, Assiut University
Other Study IDs: SDM in SLE
Record Dates: First submitted 2019-07-16; First posted 2019-07-18 (Actual); Last update posted 2023-07-19 (Actual); Status verified 2023-07

CONDITIONS: System; Lupus Erythematosus
MeSH Terms: conditions — Lupus Erythematosus, Systemic

STUDY DESIGN:
Observational Model: Other | Time Perspective: Cross-Sectional
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- SLE with corticosteroid therapy

SUMMARY:
The aim of the study is to determine the prevalence of steroid-induced diabetes mellitus (SDM) among systemic lupus erythematosus (SLE) patients and identify and assess the associated risk factors .

DETAILED DESCRIPTION:
120 SLE patients who attend the SLE and Rheumatology Clinic will be recruited into the study. All patients need to fulfil at least four criteria from the American College of Rheumatology Classification Criteria for SLE 1997(28). All patients need to be receiving corticosteroid therapy. SDM cases is defined as the development of DM after commencement of steroid treatment. Prevalent cases of SDM will also be included in the study.

Diagnosis of DM will be made according to the American Diabetes Association(29), that is fasting plasma glucose ≥ 7.0 mmol/L or HbA1c ≥ 6.5 or 2-h plasma glucose ≥ 11.1 mmol/L during an oral glucose tolerance test (OGTT). SLE patients who receive corticosteroids treatment will be screened with fasting blood sugar during out-patient clinic visit. If fasting blood glucose level is high , an additional HbA1C or OGTT will be performed.

All patients included in this study will be subjected to:

1. Full history taking: including age, sex, duration of the SLE disease , age at onset of symptoms of SLE, the progression of disease, type of corticosteroid used, dosage, duration of treatment and other types of drugs used, presence of hypertension, dyslipidemia, smoking.
2. Complete clinical examination: A standardized physical examination will be performed in all patients to measure blood pressure, waist circumference and body mass index.
3. Laboratory investigations:

   * Fasting plasma glucose.
   * HbA1c.
   * 2-h plasma glucose.
   * Total cholesterol, triglyceride, low density lipoprotein (LDL) and high density lipoprotein (HDL) levels.

ELIGIBILITY:
Inclusion criteria

* Both males and females
* Patients aged of 18-75 years.
* Clinically diagnosed as SLE patients.
* Receiving corticosteroid therapy.
* Prevalent cases of SDM with SLE.

Exclusion criteria

* SLE patients who do not receive corticosteroid therapy.
* SLE patients with other types of diabetes mellitus.

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: 120 SLE patients who attend the SLE and Rheumatology Clinic will be recruited into the study. All patients need to fulfil at least four criteria from the American College of Rheumatology Classification Criteria for SLE 1997(28). All patients need to be receiving corticosteroid therapy. SDM cases is defined as the development of DM after commencement of steroid treatment. Prevalent cases of SDM will also be included in the study.
Sampling Method: Probability Sample
Enrollment: 120 (Estimated)
Dates: Start 2022-09-01 (Actual); Primary Completion 2024-04-01 (Estimated); Study Completion 2024-04-20 (Estimated)

PRIMARY OUTCOMES:
Number of patients who developed Steroid-induced diabetes mellitus | up to 12 months post-randomization
  development of diabetes mellitus after corticosteroid therapy

SECONDARY OUTCOMES:
Number of patients who didn't develop steroid-induced diabetes mellitus | 12 months
  no development of diabetes mellitus after corticosteroid therapy

CONTACTS AND LOCATIONS:
Locations (1):
- Assiut university hospital, Asyut, Egypt